CLINICAL TRIAL: NCT01657747
Title: Whole-body Diffusion MRI for Staging, Response Prediction and Detecting Tumor Recurrence in Patients With Ovarian Cancer
Acronym: S53580
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: S53580
Record Dates: First submitted 2011-11-02; First posted 2012-08-06 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2011-09

CONDITIONS: Ovarian Carcinoma
Keywords: Ovarian carcinoma; Staging; Early treatment follow-up; Identifying tumor recurrence; Whole body diffusion-weighted MRI
MeSH Terms: conditions — Ovarian Neoplasms | interventions — gadoterate meglumine; Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Not applicable (imaging study) (No Intervention)
  Interventions: Other: Whole body diffusion-weighted MRI

INTERVENTIONS:
Other: Whole body diffusion-weighted MRI — MRI is a technique based on magnetic fields and does not require the use of ionizing radiation. Although there are no known side effects associated with MRI, a few precautions should be taken because of the 3T magnetic field. This implicates that all metal and magnetized objects must be removed from the patient before entering the MRI room. Patients with a pacemaker, a cardiac defibrillator or other implanted conductors/prostheses are for this reason not eligible for the study.
  During the whole body MRI examination, an intravenous contrast agent will be administered. In most cases, patients do not experience any discomfort and the use of this contrast agent is part of the clinical routine.
  During the whole body MRI examinations, a bowel relaxing injection (Buscopan) is also needed to reduce movement of the intestines.
  Other Names: Dotarem; Buscopan

SUMMARY:
The aim of this study is to assess whole body diffusion weighted imaging (WB-DWI) as a non-invasive method for

* accurate staging of patient suspected having ovarian cancer
* early treatment assessment
* detecting tumor recurrence

DETAILED DESCRIPTION:
1. Staging --- (PET-)CT is used nowadays to provide imaging information about the disease burden of ovarian cancer patients and a diagnostic staging laparoscopy under general anesthesia is often necessary to allow correct and accurate staging. The applicant propose an "all-in-one" imaging modality providing high quality thoracic-abdominal images without using ionizing radiation and/or radioactive material. This allows accurate assessment of operability in a minimally invasive manner.
2. Early treatment assessment --- Although response to the first administration of chemotherapy is quite reasonable, most patients show tumor recurrence and achieve increasingly poorer response rates to second- or third-line regimes. Therefore it is of major concern that a individualized prediction of chemosensitivity can be performed avoiding unnecessary toxicity from inefficient chemotherapeutic agents. A promising perspective is that the predictive data to be generated might prove to be sufficiently powerful to predict chemosensitivity early in the course of the treatment, facilitating a timely change of treatment in nonresponders. This could avoid unnecessary toxicity for patients, improving quality of life and moreover implicate considerable savings for the healthcare sector.
3. Identifying tumor recurrence --- Identifying tumor recurrence at an early stage could translate into reduction of unnecessary biopsies, cost savings and reduced morbidity associated with the biopsy procedure. But the most important issue is that early diagnosis can be life saving with respect to tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* STAGING: patients with suspected ovarian carcinoma
* EARLY TREATMENT ASSESSMENT: patients with FIGO stage IIIc or IV ovarian carcinoma who will undergo neoadjuvant chemotherapy
* IDENTIFYING TUMOR RECURRENCE: patients with a medical history of ovarian carcinoma with suspicion of recurrent ovarian cancer after a disease-free-interval of at least 6 months

Exclusion Criteria:

* patients with known contra-indications for MRI (cardiac pacemakers, cochlear implants, claustrophobic patients)will be excluded from this study.
* patients with contra-indications to gadolinium-based contrast agents (including patients with a known restricted renal function; GFR < 30 mL/min)and/or Buscopan

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validation of interpretation criteria of WB-DWI for staging and thresholding for treatment assessment in pilot study | Nov 2011 - Sep 2012 (up to 1 year)
  Validation of interpretation criteria of WB-DWI for staging and thresholding for treatment assessment in pilot study
WB-DWI for tumor characterization and staging at primary diagnosis | Nov 2011 - Nov 2015 (expected) (up to 4 years)
  The aim of this part of the study is to prospectively evaluate WB-DWI for tumor characterization and staging at primary diagnosis in comparison to CT and combined CT/diagnostic laparoscopy with the aim to assess patient operability.
WB-DWI for response assessment during and early after neoadjuvant chemotherapy | Nov 2011 - Nov 2015 (expected) (up to 4 years)
  The aim of this part of the study is to prospectively evaluate WB-DWI for (early) response assessment during and early after neoadjuvant chemotherapy in comparison to CT with the aim to predict chemotherapy induced tumor load regression and subsequent operability

SECONDARY OUTCOMES:
The prognostic value of DWI-determined imaging markers | Nov 2013 - Nov 2015 (expected) (up to 2 years)
  The aim of this part of the study is the determination of prognostic DWI-determined imaging and response markers towards patients disease free survival and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Vandecaveye, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals UZ Leuven, Gasthuisberg, Leuven, Leuven, Belgium